CLINICAL TRIAL: NCT01058330
Title: Effects of Physical Training on Bone and Muscle Quality, Muscle Strength, and Motor Coordination in Children With Neurofibromatosis Type 1
Brief Title: Effects of Physical Training on Bone and Muscle Quality, Muscle Strength, and Motor Coordination in Children With NF1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: Thrasher Research Fund (Other); University of Utah (Other)
Responsible Party: Principal Investigator, David Stevenson, MD, Assistant Professor, Division of Medical Genetics, University of Utah, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SLC00038711
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Neurofibromatosis Type 1
Keywords: Neurofibromatosis type 1; NF1
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plyometric physical training (Active Comparator): Individualized plyometric training program to increase strength, coordination, and bone density.
  Interventions: Other: Plyometric training program
- Control Group (No Intervention): This group will have no intervention

INTERVENTIONS:
Other: Plyometric training program — The intervention is a year long individualized plyometric exercise training program. Examples of plyometric activities include jumping, hopping, running, and throwing. The number of plyometric exercises will increase gradually to prevent over training to a total of five lower extremity exercises and five upper extremity exercises
  Arms: Plyometric physical training

SUMMARY:
A physical training program will improve quality of life, participation in physical activity, motor coordination, muscle strength, and bone and muscle strength in children with neurofibromatosis type 1.

DETAILED DESCRIPTION:
Disorders of the Ras pathway have significant phenotypic overlap and include Noonan syndrome, Cardiofaciocutaneous syndrome (CFC syndrome), Legius syndrome, Costello syndrome and neurofibromatosis type 1 (NF1). NF1 is one of the most common genetic disorders presenting in childhood with an incidence of 1/3000. NF1 is associated with skeletal abnormalities such as short stature, scoliosis, and long bone fracture with non-union. We recently reported that children with NF1 have abnormalities of bone and muscle architecture as evidenced by decreased bone mineral density, decreased bone strength, and low muscle mass, all of which may predispose them to fractures and scoliosis (Stevenson et al., 2005, 2007, 2009). Our preliminary data show that children with NF1 have poor motor coordination and muscle strength, potentially secondary to abnormal neuromotor learning. We hypothesize that poor motor coordination and decreased muscle strength contribute to the osteopenia in NF1. Our objective is to identify effective and non-invasive strategies to improve motor coordination, muscle strength, and bone and muscle architecture in children with disorders of the Ras pathway, in hopes of decreasing fractures and improving physical activity levels. Plyometric physical training consists of quick, high-intensity, weight-bearing movements, and is an encouraging intervention for use in these children.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill NIH clinical diagnostic criteria

Exclusion Criteria:

* Visual impairment
* Participation in a simultaneous medical intervention trial
* Orthopedic procedure within the last 6 months.
* Pregnancy
* Home location greater than 3-4 hours drive time from Shriners Hospital
* Tibial pseudarthrosis

Ages: 4 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2010-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Bone & muscle quality, DXA, pQCT, & bone ultrasound. | 1 year

SECONDARY OUTCOMES:
Motor proficiency BOT-2. Muscle strength force plate & dynamometer. Quality of life questionnaires. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David Stevenson, MD, Principal Investigator — Shriners Hospitals for Children
Locations (2):
- United States (2):
  - Shriners Hospitals for Children, Salt Lake City, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No